CLINICAL TRIAL: NCT06645938
Title: A PHASE I, RANDOMIZED, OPEN-LABEL, 2-PERIOD, 2-TREATMENT, 2-SEQUENCE, CROSSOVER, SINGLE-DOSE STUDY IN HEALTHY ADULT PARTICIPANTS TO ESTIMATE THE BIOAVAILABILITY OF AN VARIANT (HIGH HARDNESS) TABLET OF VEPDEGESTRANT (ARV-471, PF-07850327) RELATIVE TO THE REGISTRATIONAL TABLET
Brief Title: A Study to Learn How Different Tablets of the Study Medicine Vepdegestrant Are Taken up Into the Blood in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C4891038; 2024-514169-21-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-09-23; First posted 2024-10-17 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Treatment A followed by Treatment B (Experimental): Participants will receive a single 200 mg dose of vepdegestrant registrational tablet on Day 1 of Period 1 followed by a single 200 mg dose of vepdegestrant variant tablet on Day 1 of Period 2.
  Interventions: Drug: single dose of vepdegestrant as tablet formulation (Treatment A); Drug: single dose of vepdegestrant as tablet formulation (Treatment B)
- Sequence 2: Treatment B followed by Treatment A (Experimental): Participants will receive a single 200 mg dose of vepdegestrant variant tablet on Day 1 of Period 1 followed by a single 200 mg dose of vepdegestrant registrational tablet on Day 1 of Period 2.
  Interventions: Drug: single dose of vepdegestrant as tablet formulation (Treatment A); Drug: single dose of vepdegestrant as tablet formulation (Treatment B)

INTERVENTIONS:
Drug: single dose of vepdegestrant as tablet formulation (Treatment A) — Single 200 mg dose of vepdegestrant registrational (200 mg strength) tablet.
  Other Names: ARV-471, PF-07850327
Drug: single dose of vepdegestrant as tablet formulation (Treatment B) — Single 200 mg dose of vepdegestrant variant (200 mg strength) tablet.
  Other Names: ARV-471, PF-07850327

SUMMARY:
The purpose of the study is to compare the amount vepdegestrant available from two different tablet formulations under fed conditions in healthy adult participants; 200 mg vepdegestrant alternative tablet formulation compared to 200 mg vepdegestrant standard tablet formulation.

This study is seeking male or female participants of non-childbearing potential age who:

* are 18 years or older
* are healthy as decided by medical tests.
* have a Body mass index (BMI) of 16 to 32 kilogram per meter squared; and a total body weight of more than 45 kilograms (99 pounds).

All participants will be put into groups to receive one of the 2 treatments in each period. This study will consist of 2 treatment sequences:

* Sequence 1: Single 200 mg dose of vepdegestrant registrational tablet in Period 1, followed by a single 200 mg dose of vepdegestrant variant tablet in Period 2.
* Sequence 2: Single 200 mg dose of vepdegestrant variant tablet in Period 1, followed by a single 200 mg dose of vepdegestrant registrational tablet in Period 2.

Participants will be in the study for about 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male participants, and/or female participants of non-childbearing potential aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, vital signs, and standard 12-lead ECGs.
* BMI of 16-32 kg/m2; and a total body weight >45 kg (99.2 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

  * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
  * History of or active human immunodeficiency virus (HIV) infection, Hepatitis B, or Hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participants with known history of sensitivity to vepdegestrant or any of the formulation components of vepdegestrant.
* Use of any prescription or nonprescription drugs/products, dietary and herbal supplements, vitamins, grapefruit/grapefruit containing products, and Seville orange/Seville orange containing products are prohibited in this study. A washout of 7 days or 5 halflives (whichever is longer) prior to the first dose of study intervention is required. A longer washout is required for those that fall into the categories below:

  * Moderate or strong cytochrome P450 (CYP)3A inducers which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
  * Moderate or strong CYP3A inhibitors which are prohibited within 14 days or 5 half lives (whichever is longer) prior to the first dose of study intervention (unless otherwise indicated in the protocol).
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
* A positive urine drug test. A single repeat for positive drug screen may be allowed.
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Renal impairment as defined by an estimated glomerular filtration rate (eGFR) (units of mL/min/1.73 m²) in adults <60 mL/min/1.73 m² based on chronic kidney disease epidemiology (CKD-EPI) equation. Based upon participant age at screening, eGFR, is calculated using the recommended formulas to determine eligibility and to provide a baseline to quantify any subsequent kidney safety events.
* Standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTc corrected using Fridericia's formula [QTcF] >450 ms, complete left bundle branch block (LBBB), signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≥ 1.5 × upper limit of normal (ULN);
  * Total bilirubin ≥ 1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Vepdegestrant | Period 1 and 2 - pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, 120, 144, and 168 hour(s) post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Vepdegestrant | Period 1 and 2 - pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, 120, 144, and 168 hour(s) post-dose

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs). | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Clinical Laboratory Abnormalities. | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs. | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Electrocardiogram (ECG) Abnormalities. | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891038